CLINICAL TRIAL: NCT02202213
Title: Interventional, Randomised, Double-blind, Placebo Controlled, Multiple-dose Study Investigating the Safety, Tolerability, PK and PD Properties of Lu AF11167 in Patients With Schizophrenia
Brief Title: Safety and Tolerability Study of Lu AF11167 After Repeated Dosing in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15698A
Record Dates: First submitted 2014-07-25; First posted 2014-07-28 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lu AF11167 hard capsules; 0.25, 0.5 and 1 mg (Experimental): Part A: Lu AF11167 monotherapy Part B: Lu AF11167 adjunctive therapy to risperidone
  Three times daily oral dosing for 14 days.
  Interventions: Drug: Lu AF11167
- Matching placebo (Placebo Comparator): Daily oral dosing matching the experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Matching placebo
Drug: Lu AF11167
  Arms: Lu AF11167 hard capsules; 0.25, 0.5 and 1 mg

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Lu AF11167 in patients with schizophrenia following various repeated dosing regimens of Lu AF11167 (alone or as added treatment to risperidone).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged ≥18 years and ≤60 years with a body mass index (BMI) of ≥18.5 and ≤38 m2
* Primary diagnosis of schizophrenia according to DSM-IV-TR™ (codes 295.10, 295.20, 295.30, 295.90)
* Clinical Global Impression - Severity of Illness (CGI-S) score ≤4 (moderately ill) at the Screening Visit and Baseline Visit (Day -1)
* PANSS total score ≤80 at the Screening Visit and the Baseline Visit (Day -1)
* Score of 4 (moderate) of the following PANSS items at the Screening Visit and the Baseline Visit (Day -1): P7 (hostility), G8 (uncooperativeness)
* Minimal level of extrapyramidal signs, defined as a score ≤5 (moderately severe) in any of the four Clinical Global Impression of Severity (CGI-S) items of the ESRS-A; parkinsonism, akathisia, dystonia, and tardive dyskinesia at the Screening Visit and the Baseline Visit
* Willingness to be hospitalised for approximately 3 weeks after the Baseline Visit (Day -1)

Exclusion Criteria:

* The patient experienced an acute exacerbation requiring hospitalization within the last 6 months
* The patient experienced an acute exacerbation requiring increase in antipsychotic medication (with reference to drug or dose) within the last 4 weeks

Other pre-defined inclusion and exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Absolute values and changes from baseline in safety variables (Adverse events, clinical safety laboratory tests, vital signs,respiratory rate, weight, body temperature and ECG) | Screnning to day 25

SECONDARY OUTCOMES:
Columbia Suicide Severity Rating Scale (C-SSRS) | Screening to day 25

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H.Lundbeck A/S, Study Director — LundbeckClinicalTrials.com
Locations (1):
- Parexel International, Glendale, California, United States